CLINICAL TRIAL: NCT00438672
Title: Corticosteroid Injection for Common Upper Extremity Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Director of Research, Hand Service, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2003-P-000322
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-04

CONDITIONS: Lateral Elbow Pain
Keywords: lateral elbow pain; tennis elbow; pain; psychology
MeSH Terms: conditions — Tennis Elbow; Pain | interventions — Steroids; Dexamethasone; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (3):
- Dequervains (Active Comparator): The de Quervain's injection study was terminated due to difficulty with enrollment. A large percentage of patients declined, and DeQuervain's is also fairly uncommon. Therefore, the trial wasn't feasible for this diagnosis.
  Interventions: Drug: Placebo Injection; Drug: Steroid (dexamethasone) Injection
- Lateral Epicondylitis (Active Comparator)
  Interventions: Drug: Placebo Injection; Drug: Steroid (dexamethasone) Injection
- CMC Arthritis (Active Comparator): The CMC Arthritis injection study was terminated due to difficulty with enrollment. A large percentage of patients declined, and it was decided that the trial wasn't feasible for this diagnosis.
  Interventions: Drug: Placebo Injection; Drug: Steroid (dexamethasone) Injection

INTERVENTIONS:
Drug: Placebo Injection — Injection without steroid
Drug: Steroid (dexamethasone) Injection — Injection with steroid (dexamethasone)

SUMMARY:
The purpose of the study is to compare the effectiveness of a steroid injection to a placebo (inactive substance) in the treatment of lateral elbow pain, deQuervain's tendonitis, or base of the thumb carpometacarpal (CMC) arthritis. We are also trying to identify which personality factors and mindsets influence perceptions of elbow, wrist and hand pain. We hope to enroll 213 subjects in this study.

DETAILED DESCRIPTION:
Pain at the origin of the extensor carpi radialis is an extremely common problem. Most patients are between 35 and 55 years of age. This problem has been referred to as tennis elbow, but fewer than 10% of patients with this problem play tennis, and it is not a common problem among professional tennis players. The problem is most commonly called lateral epicondylitis in spite of the fact that pathology specimens show no evidence of an inflammatory process. Instead, tissue necrosis and other findings suggestive of a degenerative process are seen. Previous clinical trials have noted improvement in 80% of patients in one year, even in placebo groups, suggesting that this is a self-limited rather than a progressive disorder.

de Quervain's tenosynovitis and carpometacarpal (CMC) arthritis are also very common upper extremity problems. In de Quervain's tendonitis, inflammation in the first dorsal compartment of the wrist causes tenderness and chronic pain in the radial styloid region when forming a fist or using the thumb. CMC arthritis, most common in women 40-70, causes pain at the base of the thumb. Descriptions of the severity of this condition can range from stiffness to disability, and are associated with complaints of discomfort with pinching and gripping.

These are frustrating conditions, particularly for active people. As a consequence, varied treatments are used routinely in spite of limited scientific support. These treatments can be costly, some have risks, and all of them may reinforce the idea that there is a quick fix or miracle cure. Physicians and patients alike favor quick, direct treatments, but these are not always available. In the absence of effective treatment, the role of the physician is to encourage adaptive behaviors based upon an understanding of the nature of the illness.

Lateral elbow pain, de Quervain's tenosynovitis and CMC arthritis are extremely common and not all patients seek a physician's advice-many develop adaptive behaviors and manage well on their own. Our research unit has taken interest in studying psychological factors that may be associated with coming to the doctor and poor adaptation to symptoms and dysfunction. These are certainly a factor in the treatment of these conditions.

A condition that is extremely common; is painful and disabling; and has no clear etiology, pathophysiology, or cure represents a tempting market for products and devices claiming to offer relief. The marketing and application of these devices reinforces patient's desires for a quick fix, miracle cure. It also tends to take advantage of people with less adaptive health behaviors. Conscientious use of treatments in this setting requires strong evidence of their safety and efficacy.

Injection of corticosteroids is a common treatment for lateral elbow pain, de Quervain's tenosynovitis and CMC arthritis. Injections are delivered into the origin of the extensor carpi radialis brevis, into the first dorsal compartment of the wrist or into the trapeziometacarpal (TMC) joint, respectively. Several studies have tested the efficacy of steroid injections, including some prospective randomized trials. However, it is remarkable that only one of these have compared corticosteroid injection to placebo injection, especially in light of the fact that conditions like lateral elbow pain and de Quervain's tenosynovitis may be self-limiting. The psychological factors associated with receiving an injection may be important mediators of any treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 64 years
* onset of pain within the past 6 months
* willing to try a steroid injection in the elbow

Exclusion Criteria:

* systemic inflammatory diseases (e.g., rheumatoid arthritis)
* pregnancy
* prior steroid injection, iontophoresis treatments with corticosteroids, or surgery for their pain
* history of adverse reaction to lidocaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2003-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexamethasone Cohort: Single injection of 1 mL dexamethasone mixed with 1 mL 1% lidocaine without epinephrine
- Placebo (Lidocaine Only) Cohort: Single injection of 2 mL 1% lidocaine
Period: Overall Study
Arm/Group | Dexamethasone Cohort | Placebo (Lidocaine Only) Cohort
Started | 31 | 33
Completed | 24 | 24
Not Completed | 7 | 9
Not completed — Lost to Follow-up | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone Cohort | Placebo (Lidocaine Only) Cohort | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 31 | 62
  >=65 years | 0 | 2 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 48 (8) | 49 (10) | 49 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 12 | 15 | 27
Region of Enrollment [Number; unit: participants]
  United States | 31 | 33 | 64

OUTCOME MEASURES:

1. Primary Outcome: Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire
Description: The DASH questionnaire measures arm-specific perceived disability. It contains 30 items and is scaled between zero and 100 with higher scores indicating worse upper-extremity function.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexamethasone Cohort | Placebo (Lidocaine Only) Cohort
Number analyzed (Participants) | 24 | 24
units on a scale | 18 (20) | 13 (19)

2. Primary Outcome: Visual Analog Scale for Pain
Description: Pain is measured on a 10 cm long line that starts at 0 on the left and ends with 10 on the right. A score of 0 represents no pain at all, and a score of 10 represents the worst pain ever. The individual score is measured using a measuring rod, measuring the distance from the left border in centimeters.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexamethasone Cohort | Placebo (Lidocaine Only) Cohort
Number analyzed (Participants) | 24 | 24
units on a scale | 2.4 (2.9) | 1.7 (2.2)

ADVERSE EVENTS:
Arm/Group | Dexamethasone Cohort | Placebo (Lidocaine Only) Cohort
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/33
Other Adverse Events (participants affected / at risk) | 0/31 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No